CLINICAL TRIAL: NCT01844713
Title: Evaluation of Sun Protection Education for Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU00069552
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Unspecified Complications of Kidney Transplant; Disorder Related to Renal Transplantation
Keywords: Kidney transplant; Renal transplant; Sun protection; Skin cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: Workbook (Experimental): Distribution of the sun protection educational workbook
  Interventions: Behavioral: Workbook
- Control (No Intervention): Distribution of general skin care information

INTERVENTIONS:
Behavioral: Workbook — Subjects will read a workbook about sun protection
  Arms: Experimental: Workbook

SUMMARY:
This study is being done to evaluate the effectiveness of a Sun Protection Strategies workbook for kidney transplant recipients. Since the medication taken to preserve the kidney transplant puts kidney transplant recipients at an increased risk of developing skin cancer. The program will help people learn about how to practice effective sun protection after the transplant.

DETAILED DESCRIPTION:
Cognitive interview about the Sun Protection Strategies workbook will be performed with up to 25 kidney transplant recipients (KTR) who have participated in past surveys. A second phase of the study involves 156 KTRs that will be asked to take part in a randomized controlled trial evaluating the fully developed sun protective strategies workbook.

Kidney transplant recipients (KTRs) are at risk to develop skin cancer. Adequate sun protection after transplantation can reduce the risk of developing skin cancer. In 2006, the National Kidney Foundation (NKF) found that sun protection education delivery and content varied among transplantation centers. Clinicians rarely knew when to initiate education about skin cancer risks and prevention including timing and scope, and rarely demonstrated understanding of the importance of reminders for and repeated education of patients (National Kidney Foundation 2006).

Aims:

1. To explore culturally sensitive use of terms describing ethnic cultural perceptions of sun burning, pigment darkening after sun exposure and description of skin color by the amount of photo-protective pigment in the skin.
2. To pilot test the sun protection workbook with English speaking KTRs representing the 3 ethnic groups: White, Black and Hispanic.
3. To assess the effectiveness of an education intervention encouraging the use of sun protection strategies.
4. To explore understanding of the importance of sun protection and the KTRs confidence in their being able to practice sun protection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of kidney transplantation within the last 2-24 months
* Speaks English
* Can see to read
* Lives in the greater Chicago area and can attend two study visits
* 18-85 years old

Exclusion Criteria:

* Unable to speak English
* Cognitive impairment or neurologic disease
* Dementia or insufficient cognitive skills to follow instructions provided at a sixth grade language level
* Has had a skin cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
use of sun protection | An average of 1 year
  Subjects will complete self-report surveys of behavior prior to educational intervention and 6- 8 weeks after the educational intervention

CONTACTS AND LOCATIONS:
Overall Officials: June K. Robinson, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Faculty Foundation, Chicago, Illinois, United States